CLINICAL TRIAL: NCT00440791
Title: Evaluation of the PillCam™ Colon Capsule Endoscopy (PCCE) in the Visualization of the Colon
Status: Terminated | Type: Observational
Why Stopped: Interim analysis
Sponsor: Medtronic - MITG (Industry)
Other Study IDs: MA-54
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2007-08

CONDITIONS: Colonic Diseases
Keywords: Colon; colonic disease; capsule endoscopy; Suspected or known colonic disease
MeSH Terms: conditions — Colonic Diseases | interventions — Endoscopy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PillCam Colon capsule endoscopy

SUMMARY:
This multi-center, prospective, cohort study of 394 subjects that are indicated for standard colonoscopy due to suspected or known colonic disease examines the Given Diagnostic System and the PillCam Colon Capsule in comparison to standard colonoscopy. This study aims a. To evaluate and compare the accuracy of PillCam ™ Colon capsule endoscopy (PCCE) with standard colonoscopy. This study will evaluate the safety of PillCam ™ Colon capsule endoscopy (PCCE)

DETAILED DESCRIPTION:
The Given® Diagnostic System offers an alternative approach for endoscopic visualization of the colon using capsule endoscopy, a swallowable device which contains imagers, light sources, a power source and a RF transmitter. Advantages of the Given® Diagnostic System include the elimination of the need for conscious sedation, the minimally invasive, painless nature of the exam, and the ability to pursue normal daily activities immediately following the procedure . This multi-center prospective, cohort study will evaluate the performance of PCCE in visualizing the colon. Up to 394 subjects will participate in this study. All subjects to be enrolled will be appropriate candidates for standard colonoscopy based on their clinical indication.

Each subject will undergo PCCE. All generated PCCE RAPID videos will be reviewed by blinded PCCE reading physicians. All readers, experienced in PillCam SB, will have undergone standardized training and passed a qualification test specific to reading and interpreting PCCE videos. Training will be done by reading at least 5 cases to demonstrate proficiency in interpretation of PCCE. PCCE results will be compared with that of a colonoscopy procedure.

Following PCCE procedure, standard colonoscopy will be performed by a colonoscopist blinded to the results of the PCCE. The colonoscopist will be "unblinded" during the standard colonoscopy procedure at three locations on withdrawal of the colonoscope.

Primary Endpoint - Accuracy parameters (sensitivity, specificity, NPV, PPV) of PCCE compared to standard colonoscopy.

• Number, type and severity of adverse events with both PCCE and standard colonoscopy

ELIGIBILITY:
Inclusion criteria:

Subjects must meet one the following inclusion criteria to be eligible for enrollment into this proposed study:

Subject was referred for standard colonoscopy for one of the following reasons:

Subjects over 50 years of age with one or more of the following clinical symptoms:

rectal bleeding, hematochezia, melena, positive FOBT, recent change of bowel habits

• Any subject over 18 years of age with:

* Positive findings in the colon on a GI radiographic study (e.g., CT colonography, air-contrast barium enema, abdominal/pelvic CT scan)
* Personal history of colorectal cancer (CRC) or adenomatous colonic polyps and at least 5 years since last colonoscopy or no sooner than 3 years prior to enrollment date as long as their prior colonoscopy revealed at least one of the following high risk conditions: multiple (greater than 3)adenomas, large adenoma (greater than 1 cm) , adenomas with a villous component, adenoma with high grade dysplasia.
* Suspected or known ulcerative colitis

Exclusion criteria

The presence of any of the following will exclude a subject from study enrollment:

* Subject has dysphagia
* Subject has congestive heart failure
* Subject has renal insufficiency
* Subject is known or is suspected to suffer from intestinal obstruction.
* Subject has a cardiac pacemaker or other implanted electro medical devices.
* Subject is pregnant
* Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator.
* Subject has any condition, which precludes compliance with study and/or device instructions.
* Age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-06; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Rex, M.D., Principal Investigator — Indiana University Hospital; Glenn Eisen, M.D., Principal Investigator — Oregon Health and Science University; Rami Eliakim, MD, Principal Investigator — Rambam Health Care Campus; Jonathan Leighton, MD, Principal Investigator — Mayo Clinic; Chris Gostout, MD, Principal Investigator — Mayo Clinic; Elizabeth Rajan, MD, Principal Investigator — Mayo Clinic; Blair Lewis, MD, Principal Investigator — Private Medical Facility; S Ketover, MD, Principal Investigator — Minnesota Gastroenterology
Locations (7):
- United States (6):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Indiana University Hospital, Indianapolis, Indiana
  - Minnesota Gastroenterology, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Private Medical Facility, New York, New York
  - Oregon Health Sciences University, Portland, Oregon
- Rambam Medical Center, Haifa, Israel